CLINICAL TRIAL: NCT05588115
Title: RACE Study: Rapid, Accurate and Cost-effective Analysis of Glial Fibrillary Acid Protein Using a Hand-held Biosensor for Patient With Concussion in Acute Care and at Home Monitoring
Brief Title: Rapid, Accurate, Cost-effective Assessment of Blood Biomarkers for Diagnosis of Concussion
Acronym: RACE
Status: Recruiting | Type: Observational
Sponsor: University of Calgary (Other)
Collaborators: Foothills Medical Centre (Other)
Responsible Party: Sponsor
Other Study IDs: REB22-1015
Record Dates: First submitted 2022-10-04; First posted 2022-10-20 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Concussion, Mild
Keywords: blood biomarkers; GFAP; biosensor; concussion
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, plasma, and serum.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Concussion: Patients presenting to the ED who are diagnosed with concussion according to the ICD-10 criteria and absent of comorbidities.
- MSK: Patients presenting to the ED who are diagnosed with a muscle or skeletal injury (MSK; soft tissue damage or inflammation, fractured bone, etc.) and absent of comorbidities.

SUMMARY:
The goal of this observational study is to test if a biosensor can accurately measure a blood biomarker in adult patients presenting to the emergency department with concussion. The main questions it aims to answer are:

* Does the biosensor measure the blood biomarker of interest with the same accuracy as the current gold-standard assay technique?
* Do relationships exist between blood biomarker measurements from the biosensor and any psychological or physical symptoms of concussion?

Participants will be asked to provide blood samples at initial visit and 2-, 6-, and 12-weeks after injury while completing questionnaires at each visit, along with a brief (2 min) daily symptom inventory.

Researchers will compare the concussion group to a muscle/skeletal injury group to see if measurements from the biosensor are exclusive to concussion.

DETAILED DESCRIPTION:
BACKGROUND

It is estimated 100-300/100,000 people worldwide present to a hospital with traumatic brain injury (TBI) annually, the majority of which are classified as mild. TBI is a disruption in normal brain function caused by external biomechanical forces transmitted directly or indirectly to the head, and is a leading cause of death and disability in Canada. Approximately 1 in 450 Canadians report brain injury as their most significant injury associated with disability in the previous year. Mild traumatic brain injury (mTBI) is operationalized under clinical severity by a Glasgow Coma Scale (GCS) score of 13-15 and is often used interchangeably with concussion, though the most recent consensus definition of concussion is precluded by positive findings on standard neuroimaging techniques. Although labelled as mild with typical recovery times within two weeks of injury for adults and four weeks for youth, up to 30% of patients with concussion experience prolonged symptoms (headache, fatigue, dizziness, insomnia, depression, anxiety, poor balance, and cognitive deficits, etc.) contributing to significant functional impairment and disease burden. Furthermore, in 2016 approximately 10% of diagnosed concussions in Ontario returned to the emergency department within 14 days of injury, increasing demands on the health care system.

Lending to its identity as one of the most complex injuries to diagnose and manage, concussion currently relies on subjective measures and symptom reports as clinical indices of injury. There has been accelerated interest in addressing this limitation through research efforts working to establish objective measures of injury including advanced neuroimaging imaging techniques, machine learning of basic physiological functions (brain waves, heart rate, blood pressure, etc.), and blood biomarkers. Blood biomarkers have shown promising results regarding their ability to detect or predict severe and moderate TBI, but results in mTBI are mixed and require further investigation. Two biomarkers of brain injury - glial fibrillary acidic protein (GFAP) and ubiquitin c-terminal hydrolase L1 (UCH-L1) - were recently FDA approved to help identify necessity of a CT scan for adult mTBI patients who might have intracranial lesions. However, beyond the currently insufficient level of evidence regarding blood biomarker applications for concussion diagnosis or prognosis, an additional hurdle for future implementation in a clinical setting remains the high cost and time-consuming assay methodologies for marker detection. Single molecule array technology (SIMOA) is a fully automated immunoassay capable of biomarker detection at the femtogram level, approximately 900x more sensitive than conventional enzyme-linked immunosorbent assays. As the current gold-standard for low concentration biomarker detection, significant monetary and procedural costs may limit SIMOA's future applications for concussion biomarker detection in clinical settings. Fortunately, technological advancements are pushing the boundaries of conventional assay approaches to minimize cost and maximize efficiency, progressing towards point-of-care assay devices.

The investigators have developed a GFAP nano-biosensor capable of measuring GFAP concentrations in similar orders of magnitude as SIMOA. Briefly, the GFAP electrochemical biosensor was developed using nano-porous carbon on screen-printed electrodes with hydroxylamine (NH2OH). The nano-coated and functionalized electrodes were immobilized with monoclonal anti-human GFAP capture antibody, then blocked with bovine serum albumin. GFAP binding frequency was translated to serum concentration levels using electrochemical impedance spectroscopy (EIS). The nano-porous biosensor provided ultrasensitive GFAP detection in a wide operational range of 100 fg/mL - 10 ng/mL concentrations in the human serum. It selectively detected GFAP when tested against other biomarkers released after brain injury, and revealed a clinical sensitivity for detection of patients across TBI severities (total n=70; TBI n=26, healthy control n=44) at 84.62% (95%CI, 65.1% to 95.6%) and specificity at 61.36% (CI, 45.5% to 75.6%). The limit of detection of the GFAP biosensor was measured to be 86.6 fg/mL in serum. Additionally, our nano-biosensor demonstrated <2% intra-variation and <1% inter-variation, tackling the concern of reproducible biosensor production needed for clinical detection. This research seeks to validate the nano-biosensor in concussion patients presenting to the Emergency Department.

OBJECTIVES

Primary Aim: Establish the clinical accuracy of the GFAP nano-biosensor in patients with concussion presenting to the emergency department from diagnosis to recovery. Secondary Aim: Assess sensitivity and specificity of the GFAP nano-biosensor for identification of concussion by comparing concussion patients to musculoskeletal (MSK) injury controls. Tertiary Aim: Assess relationships between GFAP nano-biosensor concentrations and psychological (depression, anxiety), physical (headache, sleep disturbances, etc.) symptoms of concussion from diagnosis to recovery. Quaternary aim: Assess correlation between female menstrual cycle hormone concentrations (progesterone, estrogen) and GFAP nano-biosensor concentrations.

METHODS

This study has a recruitment target of 150 (equal sex representation) acute concussion patients presenting to the emergency department (ED) at foothills medical centre ages 18 through 65. Additionally, a group of 75 (equal sex representation) musculoskeletal (MSK) injury controls will be recruited from the same ED within the same age range. In a repeated measures prospective cohort design, concussion patients will complete an initial visit within 1 week of injury, then follow-up visits at 2-, 6-, and 12-weeks post-injury or until recovered. Control (MSK) patients will complete all measures at a single visit. Concussion patients who are not recovered by 12 weeks post-injury will be asked to complete questionnaires at 6 months post-injury. Study measures include clinical outcome assessments of quality of life, global health, depression, anxiety, sleep, and concussion symptoms, along with blood draws. Concussion patients will be asked to complete the post concussion symptom scale (PCSS) daily via an online link sent to them each morning to monitor recovery. For the purposes of this study, a patient will be deemed recovered if all symptoms have resolved and indicating 100% on a sliding scale that asks how recovered the patient feels from the concussion. All other questionnaires will be completed prior to initial and follow-up blood draws. Researchers will also be providing concussion patients with a QR code linked to the investigators website where patients will have access to concussion education resources to understand the injury. The two assay techniques will be compared using mean detection and distribution curves and Bland-Altman analysis. The performance of the GFAP biosensing kit in detection of uncomplicated concussion patients and monitoring their recovery will be assessed in plasma and serum. The clinical sensitivity and specificity of the GFAP biosensor in plasma and serum will be evaluated using the receiver operating characteristic (ROC) curve in comparison to SIMOA.

ELIGIBILITY:
Inclusion Criteria (concussion group):

1. diagnosed with an uncomplicated concussion according to the ICD-10 criteria with no intracranial abnormalities
2. between the ages of 18-65 years old.

Inclusion Criteria (MSK group):

1. diagnosed with any form of musculoskeletal injury in absence of comorbidities
2. between the ages of 18-65 years old

Exclusion Criteria:

1. complicated mild TBI (positive neuroimaging findings)
2. current or history of moderate or severe traumatic brain injury
3. history of neurological issue(s) (stroke, seizures, dementia, Alzheimer's, etc.) or metabolic disease(s) (diabetes, liver disease, kidney disease, cardiovascular disease, etc.)
4. greater than 7 days from injury at initial visit

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: For the exposure of interest group, adult patients (ages 18 to 65) with an uncomplicated concussion diagnosis at Foothills Medical Centre Emergency Department in Calgary Alberta will be approached to participate in this study regardless of race, ethnicity, or gender. For the control group, adult patients (ages 18 to 65) with a musculoskeletal (MSK) injury (fractured bone, connective tissue damage, etc.) at Foothills Medical Centre Emergency Department in Calgary Alberta will be approached to participate in this study regardless of race, ethnicity, or gender.
Sampling Method: Probability Sample
Enrollment: 225 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Blood serum concentrations of GFAP at initial visit | Up to 1 week following injury
  Compare serum concentrations of GFAP measured by the biosensor and the current gold-standard SIMOA technology.
Blood serum concentrations of GFAP at 2 week follow up | 2-3 weeks following injury
  Compare serum concentrations of GFAP measured by the biosensor and the current gold-standard SIMOA technology.
Blood serum concentrations of GFAP at 6 week follow up | 6-7 weeks following injury
  Compare serum concentrations of GFAP measured by the biosensor and the current gold-standard SIMOA technology.
Blood serum concentrations of GFAP at 12 week follow up | 12-13 weeks following injury
  Compare serum concentrations of GFAP measured by the biosensor and the current gold-standard SIMOA technology.
Blood plasma concentrations of GFAP at initial visit | Up to 1 week following injury
  Compare plasma concentrations of GFAP measured by the biosensor and the current gold-standard SIMOA technology.
Blood plasma concentrations of GFAP at 2 week follow up | 2-3 weeks following injury
  Compare plasma concentrations of GFAP measured by the biosensor and the current gold-standard SIMOA technology.
Blood plasma concentrations of GFAP at 6 week follow up | 6-7 weeks following injury
  Compare plasma concentrations of GFAP measured by the biosensor and the current gold-standard SIMOA technology.
Blood plasma concentrations of GFAP at 12 week follow up | 12-13 weeks following injury
  Compare plasma concentrations of GFAP measured by the biosensor and the current gold-standard SIMOA technology.

SECONDARY OUTCOMES:
Glasgow Outcome Scale Extended (GOSE) | Up to 1 week following injury
  Assesses outcomes following brain injury. Scores range from 1 to 8 with higher scores meaning better outcomes.
Glasgow Outcome Scale Extended (GOSE) | 2-3 weeks following injury
  Assesses outcomes following brain injury. Scores range from 1 to 8 with higher scores meaning better outcomes.
Glasgow Outcome Scale Extended (GOSE) | 6-7 weeks following injury
  Assesses outcomes following brain injury. Scores range from 1 to 8 with higher scores meaning better outcomes.
Glasgow Outcome Scale Extended (GOSE) | 12-13 weeks following injury
  Assesses outcomes following brain injury. Scores range from 1 to 8 with higher scores meaning better outcomes.
Glasgow Outcome Scale Extended (GOSE) | 24-25 weeks following injury
  Assesses outcomes following brain injury. Scores range from 1 to 8 with higher scores meaning better outcomes.
EuroQol - 5 Dimensions - 5 Levels (EQ-5D-5L) | Up to 1 week following injury
  Assesses general quality of life. Health state scores (not on a scale) and a visual analog scale from 0-100 with higher scores meaning better outcomes.
EuroQol - 5 Dimensions - 5 Levels (EQ-5D-5L) | 2-3 weeks following injury
  Assesses general quality of life. Health state scores (not on a scale) and a visual analog scale from 0-100 with higher scores meaning better outcomes.
EuroQol - 5 Dimensions - 5 Levels (EQ-5D-5L) | 6-7 weeks following injury
  Assesses general quality of life. Health state scores (not on a scale) and a visual analog scale from 0-100 with higher scores meaning better outcomes.
EuroQol - 5 Dimensions - 5 Levels (EQ-5D-5L) | 12-13 weeks following injury
  Assesses general quality of life. Health state scores (not on a scale) and a visual analog scale from 0-100 with higher scores meaning better outcomes.
EuroQol - 5 Dimensions - 5 Levels (EQ-5D-5L) | 24-25 weeks following injury
  Assesses general quality of life. Health state scores (not on a scale) and a visual analog scale from 0-100 with higher scores meaning better outcomes.
PROMIS Global health | Up to 1 week following injury
  Assesses mental and physical health. Scores are provided on both domains from 0 to 20 with higher scores meaning better outcomes.
PROMIS Global health | 2-3 weeks following injury
  Assesses mental and physical health. Scores are provided on both domains from 0 to 20 with higher scores meaning better outcomes.
PROMIS Global health | 6-7 weeks following injury
  Assesses mental and physical health. Scores are provided on both domains from 0 to 20 with higher scores meaning better outcomes.
PROMIS Global health | 12-13 weeks following injury
  Assesses mental and physical health. Scores are provided on both domains from 0 to 20 with higher scores meaning better outcomes.
PROMIS Global health | 24-25 weeks following injury
  Assesses mental and physical health. Scores are provided on both domains from 0 to 20 with higher scores meaning better outcomes.
Patient Health Questionnaire 9 (PHQ-9) | Up to 1 week following injury
  Assesses feelings of depression. Scores range from 0 to 27 with higher scores meaning worse outcomes.
Patient Health Questionnaire 9 (PHQ-9) | 2-3 weeks following injury
  Assesses feelings of depression. Scores range from 0 to 27 with higher scores meaning worse outcomes.
Patient Health Questionnaire 9 (PHQ-9) | 6-7 weeks following injury
  Assesses feelings of depression. Scores range from 0 to 27 with higher scores meaning worse outcomes.
Patient Health Questionnaire 9 (PHQ-9) | 12-13 weeks following injury
  Assesses feelings of depression. Scores range from 0 to 27 with higher scores meaning worse outcomes.
Patient Health Questionnaire 9 (PHQ-9) | 24-25 weeks following injury
  Assesses feelings of depression. Scores range from 0 to 27 with higher scores meaning worse outcomes.
Generalized Anxiety Disorder Questionnaire 7 (GAD-7) | Up to 1 week following injury
  Assesses feelings of anxiety. Scores range from 0 to 15 with higher scores meaning worse outcomes.
Generalized Anxiety Disorder Questionnaire 7 (GAD-7) | 2-3 weeks following injury
  Assesses feelings of anxiety. Scores range from 0 to 15 with higher scores meaning worse outcomes.
Generalized Anxiety Disorder Questionnaire 7 (GAD-7) | 6-7 weeks following injury
  Assesses feelings of anxiety. Scores range from 0 to 15 with higher scores meaning worse outcomes.
Generalized Anxiety Disorder Questionnaire 7 (GAD-7) | 12-13 weeks following injury
  Assesses feelings of anxiety. Scores range from 0 to 15 with higher scores meaning worse outcomes.
Generalized Anxiety Disorder Questionnaire 7 (GAD-7) | 24-25 weeks following injury
  Assesses feelings of anxiety. Scores range from 0 to 15 with higher scores meaning worse outcomes.
Life Event Checklist 5 (LEC-5) | Up to 1 week following injury
  Assesses exposure to potentially stressful life events. Not a scale.
Sleep and Concussion Questionnaire | Up to 1 week following injury
  Assesses sleep disturbances following concussion. Not a scale.
Sleep and Concussion Questionnaire | 2-3 weeks following injury
  Assesses sleep disturbances following concussion. Not a scale.
Sleep and Concussion Questionnaire | 6-7 weeks following injury
  Assesses sleep disturbances following concussion. Not a scale.
Sleep and Concussion Questionnaire | 12-13 weeks following injury
  Assesses sleep disturbances following concussion. Not a scale.
Sleep and Concussion Questionnaire | 24-25 weeks following injury
  Assesses sleep disturbances following concussion. Not a scale.
Pre-blood draw questionnaire | Up to 1 week following injury
  Assesses factors that may influence blood GFAP concentrations (i.e., exercise, drugs, COVID-19, etc.). Not a scale.
Pre-blood draw questionnaire | 2-3 weeks following injury
  Assesses factors that may influence blood GFAP concentrations (i.e., exercise, drugs, COVID-19, etc.). Not a scale.
Pre-blood draw questionnaire | 6-7 weeks following injury
  Assesses factors that may influence blood GFAP concentrations (i.e., exercise, drugs, COVID-19, etc.). Not a scale.
Pre-blood draw questionnaire | 12-13 weeks following injury
  Assesses factors that may influence blood GFAP concentrations (i.e., exercise, drugs, COVID-19, etc.). Not a scale.
Post Concussion Symptom Scale (PCSS) | Through study completion, on average of 2-3 weeks.
  Assesses symptoms of concussion. Scores given for total number of symptoms (0-22) and symptom severity (0-132) with

CONTACTS AND LOCATIONS:
Overall Officials: Chantel T Debert, MD, MSc, Principal Investigator — University of Calgary
Locations (1):
- Foothills Medical Centre, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cassidy JD, Carroll LJ, Peloso PM, Borg J, von Holst H, Holm L, Kraus J, Coronado VG; WHO Collaborating Centre Task Force on Mild Traumatic Brain Injury. Incidence, risk factors and prevention of mild traumatic brain injury: results of the WHO Collaborating Centre Task Force on Mild Traumatic Brain Injury. J Rehabil Med. 2004 Feb;(43 Suppl):28-60. doi: 10.1080/16501960410023732. PMID 15083870
- [Background] Najem D, Rennie K, Ribecco-Lutkiewicz M, Ly D, Haukenfrers J, Liu Q, Nzau M, Fraser DD, Bani-Yaghoub M. Traumatic brain injury: classification, models, and markers. Biochem Cell Biol. 2018 Aug;96(4):391-406. doi: 10.1139/bcb-2016-0160. Epub 2018 Jan 25. PMID 29370536
- [Background] Gordon KE, Kuhle S. Canadians Reporting Sport-Related Concussions: Increasing and Now Stabilizing. Clin J Sport Med. 2022 May 1;32(3):313-317. doi: 10.1097/JSM.0000000000000888. Epub 2020 Sep 17. PMID 32956100
- [Background] Teasdale G, Jennett B. Assessment of coma and impaired consciousness. A practical scale. Lancet. 1974 Jul 13;2(7872):81-4. doi: 10.1016/s0140-6736(74)91639-0. No abstract available. PMID 4136544
- [Background] McCrory P, Meeuwisse W, Dvorak J, Aubry M, Bailes J, Broglio S, Cantu RC, Cassidy D, Echemendia RJ, Castellani RJ, Davis GA, Ellenbogen R, Emery C, Engebretsen L, Feddermann-Demont N, Giza CC, Guskiewicz KM, Herring S, Iverson GL, Johnston KM, Kissick J, Kutcher J, Leddy JJ, Maddocks D, Makdissi M, Manley GT, McCrea M, Meehan WP, Nagahiro S, Patricios J, Putukian M, Schneider KJ, Sills A, Tator CH, Turner M, Vos PE. Consensus statement on concussion in sport-the 5th international conference on concussion in sport held in Berlin, October 2016. Br J Sports Med. 2017 Jun;51(11):838-847. doi: 10.1136/bjsports-2017-097699. Epub 2017 Apr 26. No abstract available. PMID 28446457
- [Background] McMahon P, Hricik A, Yue JK, Puccio AM, Inoue T, Lingsma HF, Beers SR, Gordon WA, Valadka AB, Manley GT, Okonkwo DO; TRACK-TBI Investigators. Symptomatology and functional outcome in mild traumatic brain injury: results from the prospective TRACK-TBI study. J Neurotrauma. 2014 Jan 1;31(1):26-33. doi: 10.1089/neu.2013.2984. Epub 2013 Oct 31. PMID 23952719
- [Background] Olesen J, Leonardi M. The burden of brain diseases in Europe. Eur J Neurol. 2003 Sep;10(5):471-7. doi: 10.1046/j.1468-1331.2003.00682.x. PMID 12940825
- [Background] Morrison L, Taylor R, Mercuri M, Thompson J. Examining Canada's return visits to the emergency department after a concussion. CJEM. 2019 Nov;21(6):784-788. doi: 10.1017/cem.2019.22. PMID 30947758
- [Background] McCrea M, Meier T, Huber D, Ptito A, Bigler E, Debert CT, Manley G, Menon D, Chen JK, Wall R, Schneider KJ, McAllister T. Role of advanced neuroimaging, fluid biomarkers and genetic testing in the assessment of sport-related concussion: a systematic review. Br J Sports Med. 2017 Jun;51(12):919-929. doi: 10.1136/bjsports-2016-097447. Epub 2017 Apr 28. PMID 28455364
- [Background] Olsson B, Lautner R, Andreasson U, Ohrfelt A, Portelius E, Bjerke M, Holtta M, Rosen C, Olsson C, Strobel G, Wu E, Dakin K, Petzold M, Blennow K, Zetterberg H. CSF and blood biomarkers for the diagnosis of Alzheimer's disease: a systematic review and meta-analysis. Lancet Neurol. 2016 Jun;15(7):673-684. doi: 10.1016/S1474-4422(16)00070-3. Epub 2016 Apr 8. PMID 27068280
- [Background] Zetterberg H, Blennow K. Fluid biomarkers for mild traumatic brain injury and related conditions. Nat Rev Neurol. 2016 Oct;12(10):563-74. doi: 10.1038/nrneurol.2016.127. Epub 2016 Sep 16. PMID 27632903
- [Background] Bazarian JJ, Biberthaler P, Welch RD, Lewis LM, Barzo P, Bogner-Flatz V, Gunnar Brolinson P, Buki A, Chen JY, Christenson RH, Hack D, Huff JS, Johar S, Jordan JD, Leidel BA, Lindner T, Ludington E, Okonkwo DO, Ornato J, Peacock WF, Schmidt K, Tyndall JA, Vossough A, Jagoda AS. Serum GFAP and UCH-L1 for prediction of absence of intracranial injuries on head CT (ALERT-TBI): a multicentre observational study. Lancet Neurol. 2018 Sep;17(9):782-789. doi: 10.1016/S1474-4422(18)30231-X. Epub 2018 Jul 24. PMID 30054151
- [Background] Kuhle J, Barro C, Andreasson U, Derfuss T, Lindberg R, Sandelius A, Liman V, Norgren N, Blennow K, Zetterberg H. Comparison of three analytical platforms for quantification of the neurofilament light chain in blood samples: ELISA, electrochemiluminescence immunoassay and Simoa. Clin Chem Lab Med. 2016 Oct 1;54(10):1655-61. doi: 10.1515/cclm-2015-1195. PMID 27071153